CLINICAL TRIAL: NCT03140189
Title: Robot- Assisted Ivor-Lewis Esophagectomy for Esophageal Cancer: Short- Term and Long Term Outcomes of a Single-Arm Phase II Trial
Brief Title: Robot-assisted IVOR-LEWIS Esophagectomy
Acronym: RAILE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hecheng Li M.D., Ph.D, Professor, Ruijin Hospital
Other Study IDs: RTS-003
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Clinical or Oncologic Benefits of Robot-assisted IVOR-LEWIS in Esophageal Cancer
Keywords: Esophageal cancer; Robotic; Ivor-Lewis esophagectomy
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Minimally invasive esophagectomy (MIE) have become increasingly popular in esophageal cancer. It is generally accepted that comparing to open resections, MIE results in decreased postoperative pain, faster recovery times, and shorter hospital stays with comparable oncologic outcomes. However, MIE poses an important challenge for established thoracic surgeons as it is a difficult technique to become skilled at with an protracted learning curve. Standard laparoscopic and thoracoscopic instruments are rigid and provide a finite freedom of movement with a two dimensional visualization of the operating field. Such a difficulty is increased even more when the Ivor-Lewis esophagectomy with an intrathoracic anastomosis is needed.

Robot- assisted surgical system has opened a new era of minimally invasive surgery. Robot- assisted surgery offers some advantages including high- definition three- dimensional visualization and 7 degrees of freedom with the use of its surgical wrists, motion scaling, and tremor filtration, allowing the surgeon to perform complex operations comfortably in the domain of urinary tract, hepatobiliary and gynecological surgery. Although a robot-assisted thoraco- laparoscopic minimally invasive esophagectomy (RAMIE) was initiated from 2003, the published experience with RAMIE remains small, especially for Ivor- Lewis approaches. The aim of this study was to investigate the short- term and long-term outcomes of RAILE to identify any clinical or oncologic benefits of RAILE in esophageal cancer.

DETAILED DESCRIPTION:
This confirmatory, nonrandomized, single-arm trial (phase II) will be conducted to evaluate short-and long-term outcomes of robot-assisted thoraco- laparoscopic minimally invasive esophagectomy for esophageal cancer. Patients will registered preoperatively. The planned sample size was 51. Preoperative endoscopic biopsy was performed in all patients to confirm the histological diagnosis of esophageal cancer. Staging workup included thorough history and physical examination, esophagogastroduodenoscopy, endoscopic ultrasonography, and integrated positron emission tomography/computed tomography scan. Patients with histologically proven malignancy were candidates for surgical procedures. Operability criteria were defined according to the National Comprehensive Cancer Network guidelines. All patients were within the American Society of Anesthesiologists (ASA) class I to III. In general, neoadjuvant chemoradiotherapy was offered to patients with T2-3 or N1-2 disease. The primary endpoint in the first stage is the short-term postoperative complications, and that in the second stage is overall survival; patients continue to be followed up for this endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven esophageal malignancy
2. All patients were within the American Society of Anesthesiologists (ASA) class I to III
3. neoadjuvant chemoradiotherapy was offered to patients with T2-3 or N1-2 disease

Exclusion Criteria:

Cancer located at the cervical esophageal Cancer located at the gastroesophageal junction history of surgery in the right thorax

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically proven malignancy were candidates for surgical procedures. Operability criteria were defined according to the National Comprehensive Cancer Network guidelines. All patients were within the American Society of Anesthesiologists (ASA) class I to III. In general, neoadjuvant chemoradiotherapy was offered to patients with T2-3 or N1-2 disease.
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2024-04-04 (Estimated)

PRIMARY OUTCOMES:
rate of major postoperative complications | 30 days after surgery

SECONDARY OUTCOMES:
rate of overall postoperative complications | 30 days after surgery
rate of 30-day mortality | 30 days after surgery
operative time | during the operation
rate of conversion | during the operation
length of hospital stay | within 30 days after surgery
rate of R0 resection | within 30 days after surgery
number of harvested lymph nodes | within 30 days after surgery
overall survival | 3 years after surgery
disease-free survival | 3 years after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Yajie Zhang, Shanghai, China

REFERENCES:
- [Background] Wee JO, Bravo-Iniguez CE, Jaklitsch MT. Early Experience of Robot-Assisted Esophagectomy With Circular End-to-End Stapled Anastomosis. Ann Thorac Surg. 2016 Jul;102(1):253-9. doi: 10.1016/j.athoracsur.2016.02.050. Epub 2016 May 4. PMID 27154153
- [Background] Park S, Hwang Y, Lee HJ, Park IK, Kim YT, Kang CH. Comparison of robot-assisted esophagectomy and thoracoscopic esophagectomy in esophageal squamous cell carcinoma. J Thorac Dis. 2016 Oct;8(10):2853-2861. doi: 10.21037/jtd.2016.10.39. PMID 27867561